CLINICAL TRIAL: NCT03820739
Title: A Cohort Study to Evaluate the Long-term Safety and Immunogenicity of the Candidate Ebola Vaccines Ad26.ZEBOV and MVA-BN®-Filo in Adults and Children
Brief Title: EBOVAC-Salone Extension
Status: Completed | Type: Observational
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: University of Sierra Leone (Other); Janssen Vaccines & Prevention B.V. (Industry); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Universiteit Antwerpen (Other)
Responsible Party: Sponsor
Other Study IDs: VAC52150EBL3005
Record Dates: First submitted 2019-01-25; First posted 2019-01-29 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-02

CONDITIONS: Ebola Virus Disease
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Subjects who received an Ebola vaccine prime vaccination in EBOVAC-Salone are eligible for enrolment in this study. Adults are defined as participants 18 years of age or older at the time of prime vaccination, and children are defined as participants aged 1 to 17 years at the time of prime vaccination in EBOVAC-Salone.
  Interventions: Other: Follow-up; Other: Blood sample collection
- Cohort 2 (offspring): Infants conceived by a female participant in EBOVAC-Salone during the 3 months following vaccination with Ad26.ZEBOV or during the 28 days following vaccination with MVA-BN®-Filo.
  Interventions: Other: Follow-up

INTERVENTIONS:
Other: Follow-up — No investigational vaccine will be administered during this study
Other: Blood sample collection — Blood sampling to assess vaccine-induced immune responses will be conducted only in cohort 1 in a subsample consisting of approximately 102 adults and 165 children (55 from each of the three paediatric age groups that were enrolled in EBOVAC-Salone: 12-17 year olds, 4-11 year olds, and 1-3 year olds).
  Groups: Cohort 1

SUMMARY:
The VAC52150EBL3005 (EBOVAC-Salone Extension) is a cohort study evaluating the long-term safety and immunogenicity of the candidate Ebola vaccines Ad26.ZEBOV and MVA-BN®-Filo in participants who were exposed to these vaccines in the VAC52150EBL3001 trial (EBOVAC-Salone, ClinicalTrials.gov Identifier: NCT02509494). No investigational vaccine will be administered during this study. The study will consist of an enrolment visit, a number of study visits and an end-of-study visit.

DETAILED DESCRIPTION:
The VAC52150EBL3005 (EBOVAC-Salone Extension) is a cohort study to evaluate the long-term safety and immunogenicity of the candidate Ebola vaccines Ad26.ZEBOV and MVA-BN®-Filo in adults and children.

Ad26.ZEBOV consists of the Janssen Vaccines & Prevention B.V. adenovirus serotype 26 (Ad26) vector expressing the glycoprotein (GP) of the Ebola virus (EBOV) Mayinga variant.

MVA-BN®-Filo consists of the Modified Vaccinia Ankara (MVA) - Bavarian Nordic (BN) vector expressing the GPs of EBOV, Sudan virus and Marburg virus and the nucleoprotein of Tai Forest virus.

These candidate Ebola vaccines are being evaluated in phase 1, 2 and 3 clinical studies, in different heterologous prime-boost regimens, in which one study vaccine is used to prime a filovirus-specific immune response and the other study vaccine is used to boost the humoral immune responses. The VAC52150EBL3001 study (EBOVAC-Salone, ClinicalTrials.gov Identifier: NCT02509494) taking place in Kambia District, Northern Sierra Leone, is a phase 3 trial with an open-label Stage 1 followed by a randomised double-blind controlled Stage 2. In Stage 1, 43 adults (aged 18 years or older) received Ad26.ZEBOV as prime followed by MVA-BN®-Filo boost vaccination at day 57. In Stage 2, approximately 400 adults and 576 children (aged 1 to 17 years - divided into three age groups; 12 to 17 years, 4 to 11 years, and 1 to 3 years), have been randomised to receive a vaccine regimen of Ad26.ZEBOV as prime and MVA-BN®-Filo as boost at day 57, or control vaccination for both prime and boost vaccination. The control used is a World Health Organisation (WHO)-prequalified Meningococcal Group A, C, W135 and Y conjugate vaccine. EBOVAC-Salone Extension has been designed to extend the total follow-up period of participants exposed to the candidate Ebola vaccines Ad26.ZEBOV and MVA-BN®-Filo in the EBOVAC-Salone study, and to follow-up infants conceived by a female participant during the 3-month period following vaccination with Ad26.ZEBOV or during the 28 day period following vaccination with MVA-BN®-Filo in EBOVAC-Salone.

STUDY OBJECTIVES

This study aims to evaluate the long-term safety and immunogenicity of the candidate Ebola vaccines Ad26.ZEBOV and MVA-BN®-Filo administered to adults and children in EBOVAC-Salone and the long-term safety of infants conceived by a female participant during the 3-month period following vaccination with Ad26.ZEBOV and the 28 day period following vaccination with MVA-BN®-Filo in EBOVAC-Salone.

Primary Objectives

* To assess the long-term safety of Ad26.ZEBOV at a dose of 5x1010 viral particles and MVA-BN®-Filo at a dose of 1x108 TCID50 (50% Tissue Culture Infective Dose) in African adults (for 5 years) and children (for 4 years).
* To assess binding antibody responses against EBOV GP, up to 5 years post-prime in adults and 4 years post-prime in children using Filovirus Animal Non-Clinical Group (FANG) enzyme-linked immunosorbent assay (ELISA).
* To assess safety, up to their fifth birthday, in infants conceived by a female participant during the 3-month period following vaccination with Ad26.ZEBOV or during the 28 day period following vaccination with MVA-BN®-Filo.

Secondary Objectives

* To assess neutralising antibody responses directed against EBOV GP as measured by a pseudovirion neutralisation assay (psVNA) at years 2, 3 and 4 post-prime in children and years 3, 4 and 5 post-prime in adults, depending on sample and assay availability.
* To evaluate the effect of previous infection with malaria, determined using validated ELISA and bead based assays, on the persistence of the humoral immune response to vaccination up to 5 years post-prime in adults and 4 years post-prime in children. The bead based assays will allow the inclusion of antigens associated with short term humoral immune responses and thus assessment of intra study exposure to malaria.

OVERVIEW OF STUDY DESIGN

This is a cohort study evaluating the long-term safety and immunogenicity of the candidate Ebola vaccines Ad26.ZEBOV and MVA-BN®-Filo in participants who were exposed to these vaccines in the EBOVAC-Salone trial. Cohort 1 will consist of participants who received an Ebola vaccine during the EBOVAC-Salone study. Adults (defined as participants 18 years of age or older at the time of the EBOVAC-Salone prime vaccination) will be followed up annually for 5 years from receipt of prime vaccination and children (defined as participants aged 1 to 17 years at the time of the EBOVAC-Salone prime vaccination) will be followed up annually for 4 years from the receipt of prime vaccination. Cohort 2 (offspring) will consist of infants conceived by a female participant in EBOVAC-Salone during the 3 months following vaccination with Ad26.ZEBOV or during the 28 days following vaccination with MVA-BN®-Filo. Offspring will be followed annually for occurrence of serious adverse events (SAEs) until their fifth birthday.

No investigational vaccine will be administered during EBOVAC-Salone Extension. The study will consist of an enrolment visit, a number of study visits and an end-of-study visit.

No study-related activities will be performed until a subject, or parent/guardian has given informed consent for their, or their child's, participation in the study. For cohort 1, enrolment into EBOVAC-Salone Extension will occur at the subject's final study visit in EBOVAC-Salone once the informed consent form (ICF) has been signed. If a subject has already completed their final study visit in EBOVAC-Salone, enrolment and baseline information will be collected at the time the participant signs the EBOVAC-Salone Extension ICF. Information from the participant's final EBOVAC-Salone study visit up to the moment of enrolment into this study will be captured retrospectively. For cohort 2, enrolment will occur once the subject's parent/guardian has signed the EBOVAC-Salone Extension ICF. Baseline information and information from birth up to the moment of enrolment into this study will be collected at the time the ICF is signed.

Study visits will take place as follows:

Cohort 1: Once yearly, on the anniversary of their prime vaccination (± 1 month), cohort 1 participants will attend the study clinic for collection of information on any SAEs since their previous visit. In a subsample of participants, blood sampling for serology assays will also be collected at each study visit.

Cohort 2: Once yearly, on their birthday (± 1 month), cohort 2 participants (offspring) will be seen at the study clinic) for collection of information on any SAEs they experienced since their previous study visit.

Between clinic visits, reminder phone calls and/or home visits will be used for retention purposes, if needed.

SUBJECT POPULATION

Cohort 1: subjects who received Ebola vaccine prime vaccination in EBOVAC-Salone are eligible for enrolment in this study.

Cohort 2: any infant conceived by a female EBOVAC-Salone participant during the 3-month period following vaccination with Ad26.ZEBOV or during the 28 day period following vaccination with MVA-BN®-Filo in EBOVAC- Salone are also eligible for this study.

DOSAGE AND ADMINISTRATION

No investigational vaccine will be administered during this study.

SAFETY EVALUATIONS

All SAEs occurring from the final EBOVAC-Salone study visit (or from birth for eligible offspring) will be collected annually as indicated in the Time and Events Schedules.

IMMUNOGENICITY EVALUATIONS

Blood sampling to assess vaccine-induced immune responses will be conducted only in cohort 1 in a subsample consisting of approximately 102 adults and 165 children (55 from each of the three paediatric age groups that were enrolled in EBOVAC-Salone: 12-17 year olds, 4-11 year olds, and 1-3 year olds). Some of the blood collected will also be used to determine previous exposure to malaria using validated ELISA and bead based assay. The immune response to malaria will be considered when evaluating the persistence of antibody response induced by the Ebola vaccines.

OTHER CLINICAL ASSESSMENTS

In both cohort 1 and cohort 2, a physical examination including vital signs will be conducted at the first study visit and at yearly visits. In cohort 2, growth measurements will also be collected. In cohort 1, a haematology assessment will be conducted in the subsample providing immunogenicity blood samples.

STATISTICAL METHODS

The primary analysis will be done when all participants have completed their final study visit or discontinued. This analysis will include all available data up to this point. No interim analyses are planned. There are no formal hypotheses tests planned for the safety data. The primary endpoint for long term safety of Ad26.ZEBOV and MVA-BN®-Filo is the occurrence of SAEs in the total vaccine cohort during the follow up period of up to 5 years (in adults) or 4 years (in children), and separately in infants in cohort 2. The primary analysis for immunogenicity will involve assessing humoral immune responses to Ad26.ZEBOV or MVA-BN®-Filo using a longitudinal design in children and adults vaccinated with Ad26.ZEBOV or MVA-BN®-Filo (cohort 1).

ELIGIBILITY:
Inclusion Criteria:

1. Must be a participant, or former participant, of the EBOVAC-Salone study, and received Ebola vaccine prime vaccination.

   or Must be an infant conceived by a female participant of EBOVAC-Salone during the 3-month period following vaccination with Ad26.ZEBOV or the 28 day period following vaccination with MVA-BN®-Filo.
2. Must consent to participate in the EBOVAC-Salone Extension study by signing (or thumbprinting, if illiterate) an ICF, indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study. If a potential participant cannot read or write, the procedures must be explained and informed consent must be witnessed by a literate third party not involved in the conduct of the study. If the potential participant is under 18 years of age, they and their parent/guardian will be informed about the study and the parent/guardian will be asked to give consent. Children aged 7 years and older will be asked to give positive assent for their participation in the study and the assent procedure must be witnessed by an adult, literate parent/guardian/third party not involved in the conduct of the study, and documented.
3. Must confirm that he/she will return to the study site for each yearly visit.

Exclusion Criteria:

1. Participants in the EBOVAC-Salone study who were allocated to the control arm receiving the WHO-prequalified Meningococcal Group A, C, W135 and Y conjugate vaccine
2. Subjects who, in the opinion of the investigator, are unlikely to adhere to the requirements of the study, or unlikely to complete follow up

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will be open to subjects who were exposed to Ad26.ZEBOV and/or MVA-BN®-Filo in the EBOVAC-Salone study.
  The study population will consist of two cohorts:
  * Cohort 1: subjects who received an Ebola vaccine prime vaccination in EBOVAC-Salone are eligible for enrolment in this study. Adults are defined as participants 18 years of age or older at the time of prime vaccination, and children are defined as participants aged 1 to 17 years at the time of prime vaccination.
  * Cohort 2 (offspring) will consist of infants conceived by a female participant in EBOVAC-Salone during the 3 months following vaccination with Ad26.ZEBOV or during the 28 days following vaccination with MVA-BN®-Filo.
Sampling Method: Non-Probability Sample
Enrollment: 653 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-07-14 (Actual)

PRIMARY OUTCOMES:
Number of Serious Adverse Events in subjects who received an Ebola vaccine prime vaccination in the EBOVAC-Salone trial. | Up to approximately 5 years in adults and 4 years in children from prime vaccination
  An SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above.
Binding antibody responses against EBOV GP using Filovirus Animal Non-Clinical Group (FANG) enzyme-linked immunosorbent assay (ELISA). | Up to approximately 5 years in adults and 4 years in children from prime vaccination
  Serum Concentration of Antibodies Binding to EBOV GP measured by Filovirus Animal Non-Clinical Group (FANG) enzyme-linked immunosorbent assay (ELISA).
Number of Serious Adverse Events, in infants conceived by an EBOVAC-Salone trial female participant during the 3-month period following vaccination with Ad26.ZEBOV or during the 28 day period following vaccination with MVA-BN®-Filo. | From birth to their fifth birthday
  An SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above.

SECONDARY OUTCOMES:
Neutralising antibody responses directed against EBOV GP as measured by a pseudovirion neutralisation assay (psVNA) | At years 2, 3 and 4 post-prime in children and years 3, 4 and 5 post-prime in adults
  psVNA: pseudovirion neutralising antibody reactivity against the EBOV GP defined as the serum titre that is able to inhibit viral infection by 50% (IC50 titer).
Effect of previous infection with malaria, determined using validated ELISA and bead based assays, on the persistence of the humoral immune response to vaccination. | Up to approximately 5 years in adults and 4 years in children from prime vaccination
  Serum concentration of malaria specific antibodies, determined using validated ELISA and bead based assays. The bead based assays will allow the inclusion of antigens associated with short term humoral immune responses and thus assessment of intra study exposure to malaria.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Watson-Jones, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Bailah Leigh, MD, Principal Investigator — University of Sierra Leone
Locations (2):
- Sierra Leone (2):
  - EBOVAC Rokupr clinic, Rokupr, Kambia
  - EBOVAC Kambia 1 clinic, Kambia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Portugal S, Tipton CM, Sohn H, Kone Y, Wang J, Li S, Skinner J, Virtaneva K, Sturdevant DE, Porcella SF, Doumbo OK, Doumbo S, Kayentao K, Ongoiba A, Traore B, Sanz I, Pierce SK, Crompton PD. Malaria-associated atypical memory B cells exhibit markedly reduced B cell receptor signaling and effector function. Elife. 2015 May 8;4:e07218. doi: 10.7554/eLife.07218. PMID 25955968
- [Result] Ryg-Cornejo V, Ioannidis LJ, Ly A, Chiu CY, Tellier J, Hill DL, Preston SP, Pellegrini M, Yu D, Nutt SL, Kallies A, Hansen DS. Severe Malaria Infections Impair Germinal Center Responses by Inhibiting T Follicular Helper Cell Differentiation. Cell Rep. 2016 Jan 5;14(1):68-81. doi: 10.1016/j.celrep.2015.12.006. Epub 2015 Dec 24. PMID 26725120
- See also: WHO. Ebola virus disease - key facts. — http://www.who.int/news-room/fact-sheets/detail/ebola-virus-disease